CLINICAL TRIAL: NCT06021665
Title: A Randomized, Double-Blind, Controlled Trial to Assess the Efficacy of a Fortetropin Supplement in Improving Symptoms of Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MYOS Corp (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20320
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Two-group, randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: Both groups and the study coordinators will be blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fortetropin Group (Experimental): The Fortetropin group will receive a 20cc size scoop with their product and will be instructed to mix 2 scoops of product with water or a milk of their choice daily.
  Interventions: Other: Fortetropin supplement
- Control Group (Placebo Comparator): The control group will receive a 50cc size scoop with their product and will be instructed to mix 2 scoops of product with water or a milk of their choice daily. The difference in scoop size is to allow for macronutrient matching of the intervention and control products.
  Interventions: Other: Cheese protein

INTERVENTIONS:
Other: Fortetropin supplement — Test Formulation: 10g serving Calories: 64.8g Carbohydrates: 0.45g Fats: 5.5g Protein: 3.38g
  Arms: Fortetropin Group
Other: Cheese protein — The cheese powder will act as the control product. Cheese powder has been chosen as it matches the macronutrient content of the test product, but without the active ingredient.
  Control Formulation: 20g serving Calories: 93g Carbohydrates: 8g Fats: 5g Protein: 3g
  Arms: Control Group

SUMMARY:
This is a hybrid, double-blind, randomized, placebo-controlled clinical trial that will last 12 weeks. Participants will be randomized into either the intervention product or control group and will consume the test product or control daily. Participants will complete study-specific and validated questionnaires at Baseline, Week 6, and Week 12, as well as blood biomarker testing for a lipid panel and high-sensitivity C-reactive protein (hs-CRP) at Baseline and Week 12.

Osteoarthritis-like symptoms, such as joint pain, inflammation, and reduced mobility will be evaluated at baseline and at each check-in. Likert scale responses will be examined from baseline to each check-in. Participant responses on product feedback will be presented as % scores. Two validated questionnaires, Western Ontario and McMaster Universities Arthritis Index (WOMAC) and the Numeric Pain Rating Scale (NPRS) will also be completed at the questionnaire time points. A full lipid panel and hs-CRP measurement will be completed via in-person blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 50-75 years of age
* Self-reporting osteoarthritis-like symptoms, experiencing 3 or more of the following symptoms: joint pain, inflammation, reduced mobility, joint swelling, and stiffness.
* Non-acute osteoarthritis, must have experienced symptoms for longer than 1 year.
* Generally healthy and don't live with any uncontrolled chronic disease
* Able to eat eggs (haven't been medically advised to avoid)
* Willing to stop eating eggs for the 12 week study

Exclusion Criteria:

* Anyone allergic or intolerant of eggs
* Anyone who has been advised to avoid eggs
* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Anyone with known severe allergic reactions.
* Women who are pregnant, breastfeeding or attempting to become pregnant
* Unwilling to follow the study protocol.
* Subjects currently enrolled in another clinical study
* Subjects having finished another clinical study within the last 4 weeks before inclusion
* Hypersensitivity, allergy, or intolerance against any compound of the test products (e. g. eggs)
* Recent implantation of a cardiac pacemaker or other active implants
* History of or present liver deficiency as defined by Quick < 70%
* History of hepatitis B, C, HIV
* Subjects who are scheduled to undergo any diagnostic intervention or hospitalization which may cause protocol deviations
* Simultaneous study participation by members of the same household
* Any diet to lose body weight
* Eating disorders or vegan diet
* Present drug abuse or alcoholism

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scoring. [Baseline to Week 12] | 12 weeks
  The WOMAC score is a widely used questionnaire-based assessment tool designed to evaluate the symptoms and functional limitations of individuals with osteoarthritis of the knee and hip joints. Patients are asked to rate their experience on a Likert scale, usually ranging from 0 to 4 or 5, where higher values indicate greater severity of symptoms or limitations.
Change in Numeric Pain Rating Scale (NPRS). [Baseline to Week 12] | 12 weeks
  The NPRS scale is a commonly used tool for assessing and quantifying pain intensity. It's a self-report scale where individuals are asked to rate their pain on a numerical scale. The scale typically ranges from 0 to 10, with 0 representing "no pain" and 10 representing "worst pain imaginable."
Changes in muscle mass perceived by participants. [Baseline to Week 12] | 12 weeks
  Survey-based assessment (0-5 scale) of participants perception of changes in muscle mass.

SECONDARY OUTCOMES:
Changes in total cholesterol. [Baseline to Week 12] | 12 weeks
  Participants will undergo blood tests to evaluate a range of parameters, including total cholesterol.
Changes in blood triglycerides. [Baseline to Week 12] | 12 weeks
  Participants will undergo blood tests to evaluate a range of parameters, including triglycerides.
Changes in High-Density Lipoprotein (HDL) cholesterol. [Baseline to Week 12] | 12 weeks
  Participants will undergo blood tests to evaluate a range of parameters, including HDL cholesterol.
Changes in Low-Density Lipoprotein (LDL) cholesterol. [Baseline to Week 12] | 12 weeks
  Participants will undergo blood tests to evaluate a range of parameters, including LDL cholesterol.
Changes in high-sensitivity C-reactive protein (hs-CRP). [Baseline to Week 12] | 12 weeks
  Participants will undergo blood tests to evaluate a range of parameters, including hs-CRP.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided